CLINICAL TRIAL: NCT06427304
Title: Cardiac Amyloidosis pRevaleNce of in OLDer Subjects Affected by Heart Failure
Acronym: ARNOLD
Status: Recruiting | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01313-42
Record Dates: First submitted 2024-04-24; First posted 2024-05-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac amyloidosis; Heart failure with left ventricular hypertrophy; Positive bone scintigraphy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tne aim purpose of this observational, multicentre and propective study is to determine the prevalence of cardiac amyloidosis in geriatric patients aged 80 years and older hospitalized within the last 12 months for heart failure with left ventricular hypertrophy (septum ≥ 12 mm) on echocardiography

DETAILED DESCRIPTION:
Patients recruitment will be curry out in 31 geriatric or cardiologic centres.

Patients will be recruited for 24 months. Each patient will participate in the study for 12 months (baseline visit, follow-up phone calls every 3 months up to 12 months i.e., at 3, 6, 9 and 12 months).

The following data will be collected at teh baseline visit: Medical history, demography, clinical data, frailty status assessed by Fried, Triage Risk Screening Tool (TRST), triggers for cardiac decompensation, biological examination, genetic testing, echocardiographic data and other data.

Bone scanning with 99mTc-DPD or 99mTc-HMDP (early or late time with SPECT will be done during hospitalization or after discharge depending on availability at the imaging centre.

The results of each examination will be evaluated to establish the existence and degree of fixation in the myocardium and to determine its distribution.

Follow-up phone s will be conducted every 3 months up to 12 months to collect hospitalizations for heart failure, hospitalizations for other cardio-vascular events, hospitalizations for non-cardiac events, admission to nursing homes or long-term care (LTC) facilities and death

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 80 years
* Hospitalised for decompensation of heart failure in the last 12 months
* Subjects with hypertrophy of the septum or left ventricle at cardiac echography (defined as ≥ 12 mm)
* Subjects able to undergo a bone scintigraphy scan
* Subjects willing to participate

Exclusion Criteria:

* Subjects refusing to participate
* Subjects admitted to palliative care unit.
* Subjects under guardianship
* Subjects with a definite diagnosis of cardiac amyloidosis

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with cardiac amyloidosis expressed by a positive bone scintigraphy.
Sampling Method: Non-Probability Sample
Enrollment: 637 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the number of patients with cardiac amyloidosis according bon scintigraphy | At inclusion

SECONDARY OUTCOMES:
Assessment of commorbidity risk according Charlson Comorbidity Index (CCI) | At inclusion
  The Charlson Comorbidity Index (CCI) assesses the level of comorbidity by considering the level of severity of 19 predefined comorbid disorders and the number of disorders present among them.
Assessment of the degree of patient dependence according Katz Index of Independence in Activities of Daily Living (ADL) | At inclusion
  Katz Index of Independence in Activities of Daily Living is an unabbreviated scale title.
  This Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Patients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Measuring cognitive impairment according Mini-Mental State Examination (MMSE) score | At inclusion
  The Mini-Mental State Examination is an unabbreviated scale title. This scale was developed as a brief screening tool to provide a quantitative evaluation of cognitive impairment and to record cognitive changes over time.
  The measure yields a total score of 30. A score of 23 or less is the generally accepted cutoff point indicating the presence of cognitive impairment. Levels of impairment have also been classified as none (24-30); mild (18-23) and severe (0-17)
Estimating the probability of neuropathic pain according "DN4 Questionnaire" | At inclusion
  This questionnaire is an unabbreviated score title, it was originally developed and validated in French (4 items of neuropathic pain). It was identified as one of the most suitable neuropathic pain screening tools for clinical use:
  * Sensitivity: Ranges from 75-98%. Proven high sensitivity for central neuropathic pain and polyneuropathies. Sensitivity is low for tigeminal neuralgia. Moderate sensitivity for detecting a neuropathic component of pain in people with chronic pain.
  * Specificity: Ranges from 37-96%.
Assessment of physical frailty according Fried scale | At inclusion
  This is an unabbreviated scale title.
  Assessment of 5 dimensions:
  * 0, 1 or 2 pathological dimensions = lack of frailty
  * 3, 4 or 5 pathological dimensions = presence of frailty
Assessment of Failty status using the Short Emergency Geriatric Assessment (SEGA) | At inclusion
  This is an unabbreviated scale title.
  * if SEGA score < ou = 8 : Not very frail
  * if it contained in the interval [9;11] : Rather frail
  * if it > ou = 12 : Very frail

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Geriatric Department, Broca hospital
Locations (36):
- France (36):
  - Geriatric Department, Broca Hospital, Paris, IIe-de-France
  - CHU Nantes, Nantes, Loire-Atlantique
  - CHU Rouen, Charles Nicole hospital, Rouen, Normandy
  - CHU Poitiers, Poitiers, Nouvelle-Aquitaine
  - CHU Montpellier, Montpellier, Occitanie
  - CHU Toulouse, Toulouse, Occitanie
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Centre Hospitalier de Carcassonne, Carcassonne
  - Centre Hospitalier Intercommunal de Castres-Mazamet, Castres
  - CHU Trousseau-Tours, Chambray-lès-Tours
  - CHU Dijon, Dijon
  - CHU Grenoble Alpes, Grenoble
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - CHU Marseille, Marseille
  - Clinique du Millénaire-Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nice, Nice
  - Hôpital Privé Gériatrique LES SOURCES-Nice, Nice
  - CHU Orléans, Orléans
  - CHU Rennes, Rennes
  - CHRU Tours-Bretonneau Hospital, Tours
  - Clinique Saint Joseph Trelaze, Trélazé
  - Médipôle Hôpital Mutualiste Villeurbanne, Villeurbanne
  - Ambroise Paré Hospital, Boulogne-Billancourt, Île-de-France Region
  - Corentin Celton Hospital, Issy-les-Moulineaux, Île-de-France Region
  - Charles Foix Hospital, Ivry-sur-Seine, Île-de-France Region
  - Emile Roux Hospital, Limeil-Brévannes, Île-de-France Region
  - GH Sud Ile-de-France, Melun, Île-de-France Region
  - Lariboisière Hospital, Paris, Île-de-France Region
  - Saint Joseph Hospital, Paris, Île-de-France Region
  - Europeen Georges Pompidou Hospital, Paris, Île-de-France Region
  - Bretonneau Hospital, Paris, Île-de-France Region